CLINICAL TRIAL: NCT03821311
Title: Investigating the Effect of Nasal High Flow Oxygen Therapy on Regional Lung Function
Acronym: INVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.376
Record Dates: First submitted 2018-12-17; First posted 2019-01-29 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Nasal High Flow; Dynamic Volumetric Computed Tomography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: It's a prospective, single-center, pilot, pathophysiological study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computed tomography examination (Experimental): Each patient will undergo a low-dose supine position chest CT scan including end-inspiratory and expiratory acquisitions, corresponding to the routine protocol for COPD patients, except that this end-inspiratory/end-expiratory CT is repeated 3 times for total of 6 CT acquisitions.
  Interventions: Radiation: Computed tomography

INTERVENTIONS:
Radiation: Computed tomography — End-inspiratory/end-expiratory CT is repeated 3 times corresponding to the 3 studied conditions: At baseline, through expiratory resistive loading using an adjustable PEP mask, and after 5 min of nasal high flow therapy at 25 L/min.
  Other Names: CT

SUMMARY:
This study aims to assess the effect of nasal high flow oxygen therapy on regional function measured by volumetric computed tomography, in patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Nasal high flow (NHF) is a non-invasive breathing therapy that is based on the delivery of heated and humidified air at flow rates that exceed peak inspiratory flow, via a large-caliber nasal cannula. It delivers a fraction of inspired oxygen (FiO2) from 21% to 100%, with a flow rate up to 60 L·min-1.

The therapy is used for a variety of disease conditions including chronic obstructive pulmonary disease (COPD). Patients with COPD frequently manifest flow limitation during resting tidal breathing, through dynamic compression of the airways, which is attributed to a loss of parenchymal tethering of the airways. In patients with severe COPD and respiratory failure, improved oxygenation and ventilation may reduce mortality. There are limited clinical data available in adult applications of NHF and on the effectiveness of NHF in patients with stable moderate or severe COPD.

The mechanisms through which NHF affects the respiratory system are still being investigated. Two of the proposed mechanisms of action of NHF therapy are the generation of 3-5 cmH20 positive airway pressure during expiration and washout of the nasopharyngeal dead space. Positive airway pressure has been shown to improve oxygenation, ventilation-perfusion matching and respiratory rates, while nasopharyngeal washout reduces the anatomical dead space and thereby improves alveolar ventilation.

Our working hypothesis is that positive nasopharyngeal pressure generated by NHF particularly during expiration can help maintain small peripheral airways patent, thereby reducing the amount of gas trapping.

Gas trapping can be quantified based on densitometric analysis of registered computerized tomography images obtained at high and low lung volumes.

ELIGIBILITY:
Inclusion Criteria:

* Stable, moderate to severe COPD, defined as follows:

Moderate: FEV1/FVC < 0.7 or lower limit of normal, and 30 < FEV1 ≤ 60 percent predicted; Severe: FEV1/FVC < 0.7 or lower limit of normal, and FEV1 ≤ 30 percent predicted

* Indication for CT imaging as part of routine workup.
* Written informed consent signed

Exclusion Criteria:

* Acute disease condition such as infection, respiratory or cardiac failure
* Persons referred to in Articles L1151-5 to L1151-8 and L1122-1-2 of the French Public Health Code: Declared pregnant, parturient or lactating, persons deprived of their liberty by judicial or administrative decision, minors, adults who are legally protected or unable to express consent, etc.
* Evolving neoplastic disease
* Patient without social security health care coverage
* Subject in an exclusion period from another study
* Any contraindication to NHF such as nasal or upper airway bleeding, secretion, tumor, recent surgery; cervical, nasal or skull fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Gas trapping (expressed as percent total lung volume) | 30 minutes

SECONDARY OUTCOMES:
Regional lung ventilation distribution | 30 minutes
  Regional change in attenuation between end-expiration and end-inspiration, based on CT image
Coefficient of variation of regional lung ventilation | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Stubbing DG, Pengelly LD, Morse JL, Jones NL. Pulmonary mechanics during exercise in subjects with chronic airflow obstruction. J Appl Physiol Respir Environ Exerc Physiol. 1980 Sep;49(3):511-5. doi: 10.1152/jappl.1980.49.3.511. PMID 7204175
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Pisani L, Vega ML. Use of Nasal High Flow in Stable COPD: Rationale and Physiology. COPD. 2017 Jun;14(3):346-350. doi: 10.1080/15412555.2017.1315715. Epub 2017 May 1. PMID 28459282
- [Background] Curley GF, Laffy JG, Zhang H, Slutsky AS. Noninvasive respiratory support for acute respiratory failure-high flow nasal cannula oxygen or non-invasive ventilation? J Thorac Dis. 2015 Jul;7(7):1092-7. doi: 10.3978/j.issn.2072-1439.2015.07.18. No abstract available. PMID 26380720
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Background] Spahija J, de Marchie M, Grassino A. Effects of imposed pursed-lips breathing on respiratory mechanics and dyspnea at rest and during exercise in COPD. Chest. 2005 Aug;128(2):640-50. doi: 10.1378/chest.128.2.640. PMID 16100149
- [Background] O'Donnell DE, Sanii R, Anthonisen NR, Younes M. Expiratory resistive loading in patients with severe chronic air-flow limitation. An evaluation of ventilatory mechanics and compensatory responses. Am Rev Respir Dis. 1987 Jul;136(1):102-7. doi: 10.1164/ajrccm/136.1.102. PMID 3605825
- [Background] Mueller RE, Petty TL, Filley GF. Ventilation and arterial blood gas changes induced by pursed lips breathing. J Appl Physiol. 1970 Jun;28(6):784-9. doi: 10.1152/jappl.1970.28.6.784. No abstract available. PMID 5419502
- [Background] Galban CJ, Han MK, Boes JL, Chughtai KA, Meyer CR, Johnson TD, Galban S, Rehemtulla A, Kazerooni EA, Martinez FJ, Ross BD. Computed tomography-based biomarker provides unique signature for diagnosis of COPD phenotypes and disease progression. Nat Med. 2012 Nov;18(11):1711-5. doi: 10.1038/nm.2971. Epub 2012 Oct 7. PMID 23042237
- [Background] Fricke K, Tatkov S, Domanski U, Franke KJ, Nilius G, Schneider H. Nasal high flow reduces hypercapnia by clearance of anatomical dead space in a COPD patient. Respir Med Case Rep. 2016 Aug 26;19:115-7. doi: 10.1016/j.rmcr.2016.08.010. eCollection 2016. PMID 27668173
- [Background] Kybic J, Unser M. Fast parametric elastic image registration. IEEE Trans Image Process. 2003;12(11):1427-42. doi: 10.1109/TIP.2003.813139. PMID 18244700
- [Background] Gibson GJ, Loddenkemper R, Lundback B, Sibille Y. Respiratory health and disease in Europe: the new European Lung White Book. Eur Respir J. 2013 Sep;42(3):559-63. doi: 10.1183/09031936.00105513. No abstract available. PMID 24000245
- [Derived] Cohen JG, Broche L, Machichi M, Ferretti GR, Tamisier R, Pepin JL, Bayat S. Nasal High Flow at 25 L/min or Expiratory Resistive Load Do Not Improve Regional Lung Function in Patients With COPD: A Functional CT Imaging Study. Front Physiol. 2021 Jun 10;12:683316. doi: 10.3389/fphys.2021.683316. eCollection 2021. PMID 34177626